CLINICAL TRIAL: NCT04596020
Title: Can Blood Flow Restriction Therapy Improve Strength and Muscle Cross-Sectional Area for Shoulder External Rotators Better Than Exercise Alone?
Brief Title: Can Blood Flow Restriction Therapy Improve Strength and Cross-Sectional Area for Shoulder External Rotators Better Than Exercise Alone?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: George Fox University (Other)
Responsible Party: Principal Investigator, Jason Brumitt, Associate Professor of Physical Therapy, George Fox University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2183025
Record Dates: First submitted 2020-10-08; First posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Can Blood Flow Restriction Therapy Augments Strength Gains in the Rotator Cuff; Muscle Weakness
Keywords: blood flow restriction; shoulder
MeSH Terms: conditions — Muscle Weakness | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The assessors will not be aware of group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blood Flow Restriction Group (Experimental): This group will perform 2 lower extremity exercises (sitting unilateral knee extension, standing unilateral knee curl) under occlusion (i.e., BFR) for 4 sets (30/15/15/15 reps) each followed by 2 shoulder exercises (scaption and sidelying external rotation) 3 sets x 15 reps each. Exercises will be performed at 30% of 1RM.
  Interventions: Other: Blood Flow Restriction Group (exercise with blood flow restriction using a Delfi unit)
- Non-Blood Flow Restriction Group (Active Comparator): This group will perform the same exercises for the same volume without the use of BFR.
  Interventions: Other: Blood Flow Restriction Group (exercise with blood flow restriction using a Delfi unit)

INTERVENTIONS:
Other: Blood Flow Restriction Group (exercise with blood flow restriction using a Delfi unit) — Each group performs the same 4 exercises The BFR group will utilize the Delfi BFR unit
  Other Names: Non-Blood Flow Restriction Group (exercise without blood flow restriction)

SUMMARY:
This 8-week study will investigate whether the application of blood flow restriction (BFR) therapy augments rotator cuff strength in untrained individuals. This is a RCT with subjects randomized to a BFR or non-BFR group. Both groups will do the same training program: 1) first sitting unilateral knee extension and standing unilateral knee curls (w/ or w/o BFR; 4 sets, 30/15/15/15 reps) and 2) scaption and sidelying external rotation (no BFR for either group; 3 sets x 15 reps each).

DETAILED DESCRIPTION:
This 8-week study will investigate whether the application of blood flow restriction (BFR) therapy augments rotator cuff strength in untrained individuals. This is a RCT with subjects randomized to a BFR or a non-BFR group. Both groups will perform the same training program 2 times a week over 8 weeks with one group performing the lower extremity exercises under occlusion (i.e., BFR applied to the proximal thigh of the dominant leg).

Prior to starting the study the subjects will have their strength assessed by a blinded physical therapist using a hand held dynamometer. The muscles assessed will be the: quadriceps, the hamstrings, the supraspinatus, and the external rotators of the shoulder. Another blinded physical therapist will assess the cross-sectional area of the quadriceps and the supraspinatus tendon using ultrasonography. These tests will be repeated at the conclusion of the study.

Subjects' training weight will be 30% of their 1 repetition max (1RM). 1RM will be determined using hand held dumbbells for the shoulder exercises and machines (knee extension, knee curl machines) for the lower extremity exercises.

Subjects will be randomized to either the BFR or non-BFR group. Subjects in the BFR group will perform the lower extremity exercises under occlusion (i.e., BFR applied to the proximal thigh of the dominant lower extremity). Both groups will perform 4 sets of each lower extremity exercise for 30/15/15/15 reps. After completing the lower extremity exercises the subjects will perform the shoulder exercises (scaption, sidelying external rotation) for 3 sets of 15 repetitions each. The shoulder exercises will not be performed with BFR in either group.

ELIGIBILITY:
Inclusion Criteria:

• Male or female subjects aged 18 and over

Exclusion Criteria:

* Current neck, shoulder (or general upper extremity), and/or thoracic spine pathology;
* Shoulder surgery (or general upper extremity surgery) during the prior 6-month time period;
* Current lower extremity injury and/or having had a lower extremity surgery during the prior 6-month time period;
* Cervical/thoracic spine surgery during the prior 1-year;
* Subject having 1 or more contraindications for BFR training;
* Under the age of 18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-10-10 (Actual); Primary Completion 2020-12-07 (Estimated); Study Completion 2020-12-07 (Estimated)

PRIMARY OUTCOMES:
Strength Assessment | Change in Baseline Strength (Newtons) at 8 weeks
  Strength will be assessed using a hand held dynamometer and traditional manual muscle test positions
Ultrasonography | Change in Baseline Cross-Sectional Area of the Quadriceps (specifically Rectus Femoris) and the Supraspinatus tendon at 8 Weeks
  Diagnostic ultrasound will be used to measure the cross-sectional area of the quadriceps (specifically the Rectus Femoris) and the tendon of the supraspinatus

CONTACTS AND LOCATIONS:
Overall Officials: Jason Brumitt, PhD, Principal Investigator — College of Physical Therapy, George Fox University
Locations (1):
- George Fox University, Newberg, Oregon, United States

IPD SHARING:
Plan to Share IPD: No